CLINICAL TRIAL: NCT03504306
Title: Validation of Ventriject Determined Maximal Oxygen Uptake
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Prof. Jørn Wulff Helge, University of Copenhagen
Other Study IDs: Ventriject1
Record Dates: First submitted 2018-03-15; First posted 2018-04-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples for testing blood values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ventriject validation — comparing measurements from echocardiography, echoseismography to measurements of maximal oxygen uptake

SUMMARY:
This study aims to validate the use of the Ventriject product to estimate VO2 max, through a non-physically active test using ECG, echoseismography and echosonography.

DETAILED DESCRIPTION:
this study will be composed of the following tests:

* blood sample for measurement of blood values
* blood pressure measurement to rule out risks affiliated with maximal effort testing
* DXA body composition scanning
* Measurement on ECG, echosonography and echoseismography with accelerometer, microphone and ECG wires
* Measurements with phone (iPhone)
* VO2 max assessment by maximal oxygen uptake testing on a training bike, using online oxygenmeasurement equipment
* Hand-grip strength assessment

ELIGIBILITY:
Inclusion Criteria:

- healthy adults between 18 and 45 years of age

Exclusion Criteria:

* current or previous cardiovascular disease
* chronic use of medicine
* pregnancy
* illnesses which prohibits the testing of maximal oxygen uptake

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 50/50 gender composition, meaning uptake of participants of a gender will end when the group reaches 50 participants
Study Population: healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Comparing how well the Ventriject software can estimate VO2 max | 4 months data collection, although cross sectional
  VO2 max tested on bike with online software Ventriject will estimate VO2max based on ECG, echoseismography and echosonography obtained at rest

SECONDARY OUTCOMES:
comparing how well the measurements from the mobile phone test compare to the same measurements with accelerometer and echosonography | 4 months data collection, although cross sectional
  comparison of ECG, echoseismography and echosonography obtained at rest to a measurement of movement (caused by heart contraction) by mobile phone, also at rest

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, Prof., Principal Investigator — jhelge@sund.ku
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPD is possible if the following terms are met:
  1. Identification of the study participant is in no way achieveable from the requested data
  2. The participant declares interest in their data being shared through IPD